CLINICAL TRIAL: NCT00831298
Title: Assessment of Sleep Disturbance in Alzheimer Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 08-PP-07
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Alzheimer Disease
Keywords: alzheimer disease; sleep disturbance; apathy; memory loss
MeSH Terms: conditions — Alzheimer Disease; Parasomnias; Lethargy; Memory Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Behavioral Questionnaire Sleep Recordings Genetic analysis
  Interventions: Other: Analysis of sleep disturbance

INTERVENTIONS:
Other: Analysis of sleep disturbance — Behavioral Questionnaire Sleep Recordings Genetic analysis

SUMMARY:
The purpose of this study is to study circadian rhythms, or daily cycles of sleep, wake, and activity. The investigators hope to learn how disturbed sleep in Alzheimer's Disease relates to changes in activity cycles, and how sleep disturbances may affect your daytime alertness.

This project selects patients suffering from memory problems, or voluntary to be in our Control Group. There are three parts to this study: Sleep Diaries, Behavioral Questionnaire, and Activity Recordings

ELIGIBILITY:
Inclusion Criteria:

* alzheimer disease
* MMSE > 20
* over 65 years old

Exclusion Criteria:

* new psychotropic drug treatment
* patient unable to do neuropsychologic tests

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
assessment of apathy | at day 0, just after inclusion

SECONDARY OUTCOMES:
assessment of sleep disturbance | during a week, between day 0 and day 7
determine a genetic relationship between sleep disturbance and alzheimer disease | after all genetic analyses of the study

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROBERT, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Centre Mémoire de Ressources et de Recherche, CHU de Nice, Nice, France